CLINICAL TRIAL: NCT00203190
Title: A Single-Center, Randomized, Double-Blind, Placebo Controlled Trial Examining the Safety and Efficacy of Topiramate in the Treatment of Subjects With Episodic or Chronic Cluster Headache.
Brief Title: A Double-Blind, Placebo-Controlled Study Examining the Use of Topiramate in the Treatment of Cluster Headache
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SDS/TOP-CL/01/CAPSS-322; 080-19000-H56501
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
Topiramate is a medication that has been approved by the Food and Drug Administration (FDA) for the treatment of patients with seizures. The trade name for this drug is Topamax®. Topiramate has not been approved by the FDA for the treatment of cluster headache and is experimental for the purposes of this research study. If a subject participates in this study, he/she will increase his/her dose of topiramate rapidly in the first few weeks to try to stop the cluster attacks and then will continue on a maintenance dose of topiramate in order to determine if it can prevent attacks from occurring during that cluster period. We believe that this will lead not only to a faster but a more complete remission of the cluster period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 and 65 with a diagnosis of cluster headache (episodic or chronic) as defined by the International Classification of Headache Disorders (2nd edition)
* Subjects must have a lifetime prevalence of at least 2 prior cluster cycles.
* Subjects must experience one or more attacks/ day during baseline period
* Subjects must have a typical cluster period lasting at least 8 weeks. Subjects must present in active cluster period and the expected remaining duration of the cluster cycle must be at least 8 weeks from Baseline visit.
* Subjects with other headache types are eligible provided the subject is able to differentiate these headaches from cluster headaches.
* Subject is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator), if female of child-bearing potential
* Subject has negative urine pregnancy test prior to study entry, if female of child-bearing potential
* Subject is able to understand and comply with all study requirements
* Subject provides written informed consent prior to any screening procedures being conducted

Exclusion Criteria:

* Women who are pregnant or lactating
* Subjects who, in the investigators opinion, have a history or have evidence of a medical or psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial
* Subjects who require a change in medication or existing regimen of medication for the prophylaxis of cluster in the 4 weeks prior to Baseline visit and for the duration of the trial
* Subjects who have cluster headaches that typically exceed 4 hours
* Subjects who have used the following medications/ treatments from four weeks prior to Baseline visit: corticosteroids and nerve blocks.
* Subjects using any drug which might interact adversely with, or interfere with the action of, the study medication (e.g., carbonic anhydrase inhibitors)
* Subjects who have failed an adequate trial of topiramate for cluster headaches due to lack of efficacy or adverse events, as determined by the investigator
* Subjects with a history of nephrolithiasis.
* Subjects who are allergic to or have shown hypersensitivity topiramate or agents similar to topiramate
* Subjects who abuse opioids as determined by investigator
* Subjects with a history of significant drug or alcohol abuse within the past year
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-09; Study Completion 2006-06

PRIMARY OUTCOMES:
Change in the average daily frequency of moderate or severe attacks between baseline period to the period of day 14 to 56.

SECONDARY OUTCOMES:
Change in the average daily frequency of any attacks from the baseline period through the entire treatment period.
Change in the average daily duration of any attacks from the baseline period through the entire treatment period.
Change in the average daily attack severity from baseline period through the entire treatment period.
Change in the average daily frequency of any attacks from the baseline period to each week during the treatment period.
Change in the average daily duration of any attacks from the baseline period to each week during the treatment period.
Change in the average daily attack severity from the baseline period to each week during the treatment period.
Time to the first week from the baseline period with a 50% reduction in average daily frequency of moderate or severe attacks.
Change in use of acute and rescue medications from the baseline period through the entire treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: William B Young, MD, Principal Investigator — Thomas Jefferson University, Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States